CLINICAL TRIAL: NCT00004553
Title: Diagnosis of Neuromuscular Disorders With Specialized Electromyographic Studies
Brief Title: Electromyography to Diagnose Neuromuscular Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000072; 00-N-0072
Record Dates: First submitted 2000-02-04; First posted 2000-02-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Healthy; Neuromuscular Disease; Postpoliomyelitis Syndrome
Keywords: Single Fiber EMG; Macro-EMG; Myasthenia; Post-Polio Syndrome; Neuromuscular Transmission; Motor Dysfunction; Neuromuscular Disorder
MeSH Terms: conditions — Neuromuscular Diseases; Postpoliomyelitis Syndrome; Neurologic Manifestations | interventions — Neurofeedback

INTERVENTIONS:
Procedure: Electromyography

SUMMARY:
This study will investigate problems with muscle weakness and control using electromyography-a test of nerve-muscle cell communication. Advanced techniques called single fiber electromyography and macro-electromyography, which evaluate individual muscle fibers, will be used. Besides aiding in diagnosis, these tests provide information about disease progression that may be useful in guiding therapy.

Adult patients with suspected neurological disorders of muscle control and weakness may be eligible for this study. Normal volunteers may also participate. For the electromyography procedure, a special needle is inserted into a muscle. The patient will slightly tense the muscle and maintain the tension while electrical signals from the muscle fibers are being recorded. The electrical signals are played through a loudspeaker, providing feedback to help the patient tense the muscle the appropriate amount. The test, which is usually done for only one muscle, takes 1 to 2 hours. If needed, short breaks can be taken.

If the patient cannot maintain tension in the muscle for the entire test period, a nerve will be stimulated to activate the muscle. A thin needle is inserted near the nerve, and a series of small electrical shocks are given to activate a nerve fiber. The electromyography needle is inserted into the muscle to measure the response, as described above.

A neurologist receiving specialized training in clinical neurophysiology will do the electromyography procedure under the direct supervision of an experienced neurologist.

DETAILED DESCRIPTION:
This is a training protocol to enable fellows in clinical neurophysiology to learn and perform technically advanced electrodiagnostic studies, such as single fiber EMG and macro EMG, on patients with neuromuscular diseases.

ELIGIBILITY:
INCLUSION CRITERIA:

Adult patients with weakness or motor dysfunction: 8/year.

Normal volunteers, adults: 2/year.

EXCLUSION CRITERIA:

Anticoagulation or uncorrected bleeding disorder.

Children are not optimal subjects for fellows undergoing training in these techniques and will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2000-02; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Sanders DB, Stalberg EV. AAEM minimonograph #25: single-fiber electromyography. Muscle Nerve. 1996 Sep;19(9):1069-83. doi: 10.1002/(SICI)1097-4598(199609)19:93.0.CO;2-Y. PMID 8761262
- [Background] Grimby G, Stalberg E, Sandberg A, Sunnerhagen KS. An 8-year longitudinal study of muscle strength, muscle fiber size, and dynamic electromyogram in individuals with late polio. Muscle Nerve. 1998 Nov;21(11):1428-37. doi: 10.1002/(sici)1097-4598(199811)21:113.0.co;2-x. PMID 9771666